CLINICAL TRIAL: NCT00612235
Title: Comparison of Different Antiepileptic Drug Monotherapies for the Occurrence of Premenstrual Dysphoric Disorder Among Women With Epilepsy
Brief Title: Premenstrual Dysphoric Disorder and Antiepileptic Drugs
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Newton-Wellesley Hospital (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Herzog, Professor of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2007P000357
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-01

CONDITIONS: Epilepsy
Keywords: epilepsy; lamotrigine; levetiracetam; carbamazepine; phenytoin; lamictal; keppra; tegretol; carbatrol; dilantin
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine; Levetiracetam; Carbamazepine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Lamotrigine Monotherapy: Lamotrigine Monotherapy
  Interventions: Drug: Lamotrigine
- Levetiracetam Monotherapy: Levetiracetam Monotherapy
  Interventions: Drug: Levetiracetam
- Carbamazepine Monotherapy: Carbamazepine Monotherapy
  Interventions: Drug: Carbamazepine
- Normal control (no epilepsy): Normal control (no epilepsy)
  Interventions: Other: No Intervention

INTERVENTIONS:
Drug: Lamotrigine — Subjects had at least 3 months on a stable dosage of lamotrigine monotherapy.
  Other Names: Lamictal
  Groups: Lamotrigine Monotherapy
Drug: Levetiracetam — Subjects had at least 3 months on a stable dosage of levetiracetam monotherapy.
  Other Names: Keppra
  Groups: Levetiracetam Monotherapy
Drug: Carbamazepine — Subjects had at least 3 months on a stable dosage of carbamazepine monotherapy.
  Other Names: Tegretol
  Groups: Carbamazepine Monotherapy
Other: No Intervention — No intervention was given
  Groups: Normal control (no epilepsy)

SUMMARY:
This study is being done to determine if there are differences in mood during the menstrual cycle among women with epilepsy who take various different antiepileptic drugs and women without epilepsy.

DETAILED DESCRIPTION:
Participants will be given informed consent during the initial study visit. We will gather information about their seizure disorder and medications and provide them with instructions and a form that they will complete daily for two months (two menstrual cycles). During the third week of each menstrual cycle, they will be asked to return once to provide a blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Women with epilepsy, 18-45 years of age. Women will be on one of 4 established (≥ 3 months) AED monotherapies: LTG, CBZ, PHT or LEV and with documented therapeutic range serum AED level during the year prior to enrollment.
* Normal Control women, 18-45 years of age, in good general health by history

Exclusion Criteria:

* Concomitant use of prescribed or OTC reproductive hormones
* Concomitant use of antidepressant and anxiolytic medications such as SSRIs, bupropion, tricyclics, benzodiazepines

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Three regional epilepsy centers
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Herzog, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts

REFERENCES:
- [Background] Herzog AG, Smithson SD, Fowler KM, Krishnamurthy KB, Sundstrom D, Kalayjian LA, Heck CN, Oviedo S, Correl-Leyva G, Garcia E, Gleason KA, Dworetzky BA. Premenstrual dysphoric disorder in women with epilepsy: relationships to potential epileptic, antiepileptic drug, and reproductive endocrine factors. Epilepsy Behav. 2011 Aug;21(4):391-6. doi: 10.1016/j.yebeh.2011.05.024. Epub 2011 Jul 2. PMID 21724471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 3 participating sites enrolled 60 women with epilepsy, 20 in each of the 3 antiepileptic drug groups, and 20 normal controls between 4/1/2008 and 3/31/2010. All of the women met inclusion and exclusion criteria. No enrolled subject was excluded after enrollment.
Pre-assignment Details: Since the original conceptualization of the study, phenytoin use declined among women with epilepsy in the general population to the point that we did not identify a sufficient base population in our initial screen to proceed with enrollment of this group and the decision was made at the start of the study to exclude this drug group.
Groups:
- 1 Lamotrigine Monotherapy: Women with Epilepsy on Lamotrigine Monotherapy
- 2 Levetiracetam Monotherapy: Women with Epilepsy on Levetiracetam Monotherapy
- 3 Carbamazepine Monotherapy: Women with Epilepsy on Carbamazepine Monotherapy
- 5 Normal Control: Normal Control Women(no epilepsy)
Period: Overall Study
Arm/Group | 1 Lamotrigine Monotherapy | 2 Levetiracetam Monotherapy | 3 Carbamazepine Monotherapy | 5 Normal Control
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Women with epilepsy on antiepileptic drug monotherapies and normal controls. There was no difference in the number who started and completed.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Lamotrigine Monotherapy | 2 Levetiracetam Monotherapy | 3 Carbamazepine Monotherapy | 5 Normal Control | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 20 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.44 (8.06) | 33.08 (7.57) | 29.93 (8.74) | 31.79 (8.21) | 31.75 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 20 | 20 | 80
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: To Determine if the Frequency of Premenstrual Dysphoric Disorder Differs Among Various Antiepileptic Drug Monotherapies.
Description: Proportion of women who meet the Endicott Daily Record of Severity of Problems (DRSP) criteria for PMDD for two consecutive menstrual cycles in women with epilepsy and the control group (no epilepsy). To meet PMDD designation, women must have reached the PMDD criteria for both menstrual cycles. The less stringent threshold for PMDD designation referred to (1) having more severe symptoms during the premenstrual phase than during the midfollicular phase regardless of whether the midfollicular symptom scores exceeded the Endicott cutoff and (2) meeting the other three Endicott criteria
Time Frame: Assessment of PMDD Designation after two consecutive menstrual cycles
Measure: Count of Participants; unit: Participants
Arm/Group | 3 Carbamazepine Monotherapy | 2 Levetiracetam Monotherapy | 1 Lamotrigine Monotherapy
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Endicott PMDD Designation | 0 | 0 | 0
  Less Stringent Threshold for PMDD Designation | 2 | 2 | 2
  No PMDD Designation | 18 | 18 | 18

2. Primary Outcome: Proportion of Women With PMDD in WWE and the Control Group
Description: as for outcome 1
Time Frame: Assessment of PMDD Designation after two consecutive menstrual cycles
Measure: Count of Participants; unit: Participants
Groups:
- Women With Epilepsy: Women with Epilepsy
- Control Group: Women without Epilepsy
Arm/Group | Women With Epilepsy | Control Group
Number analyzed (Participants) | 60 | 20
Participants
  Endicott PMDD Designation | 0 | 0
  Less Stringent Threshold for PMDD Designation | 6 | 2
  No PMDD Designation | 54 | 18

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Lamotrigine: Women with Epilepsy on Lamotrigine Monotherapy
- Levetiracetam: Women with Epilepsy on Levetiracetam Monotherapy
- Carbamazepine: Women with Epilepsy on Carbamazepine Monotherapy
- Control: Normal control (no epilepsy)
Arm/Group | Lamotrigine | Levetiracetam | Carbamazepine | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No